CLINICAL TRIAL: NCT06232551
Title: eVTE (Electronic Venous Thromboembolism): A Cluster, Randomized, Step-wedge Type II Hybrid Study of an Alert Recommending Extended Duration Thromboprophylaxis for At-risk Discharging Medical Patients to Prevent VTE.
Brief Title: Alerting Providers at Patient Hospital Discharge to Consider Prescribing Rivaroxaban to Reduce Venous Thromboembolism
Acronym: eVTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scott C. Woller, MD (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Scott C. Woller, MD, Physician, thrombosis service, Intermountain Medical Center, Intermountain Health Care, Inc.
Organization: Intermountain Health Care, Inc. (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 1052468
Record Dates: First submitted 2024-01-18; First posted 2024-01-30 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Venous Thromboembolic Disease; Pulmonary Embolism and Thrombosis; Deep Vein Thrombosis; Hospitalism
Keywords: post-discharge; extended duration thromboprophylaxis; rivaroxaban; direct oral anticoagulant; medical patient
MeSH Terms: conditions — Pulmonary Embolism; Thrombosis; Venous Thrombosis | interventions — Electronic Health Records; Caffeine

STUDY DESIGN:
Intervention Model Description: Cluster-randomized, Type II hybrid implementation effectiveness study with step-wedge implementation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- At-risk patients for which an alert is sent during the intervention phase (Experimental): Patients found to be at an increased risk for VTE but a low risk for bleeding (based upon eVTE risk assessment), thereby meeting criteria for alerting during the intervention phase
  Interventions: Other: EHR (electronic health record) alert
- At-risk patients during the baseline phase (Active Comparator): Patients found to be at an increased risk for VTE but a low risk for bleeding (based upon eVTE risk assessment), and who meet criteria for alerting, but for whom no alert is sent during the baseline phase
  Interventions: Other: No EHR (electronic health record) alert

INTERVENTIONS:
Other: EHR (electronic health record) alert — Pop-up alert that informs the discharging clinician that the patient meets criteria to be considered for extended duration thromboprophylaxis
  Arms: At-risk patients for which an alert is sent during the intervention phase
Other: No EHR (electronic health record) alert — During the baseline phase while risk is assessed and stored, no alerting occurs
  Arms: At-risk patients during the baseline phase

SUMMARY:
A new algorithm derived from only patient age and components of the complete blood count and basic metabolic panel can identify patients discharged from the hospital who may benefit from a blood thinner (called rivaroxaban) to decrease their risk of blood clots, and for whom the risk of bleeding is minimal.

The purpose of this study is to evaluate the use of a pop-up alert, which will be seen by clinicians when a discharging patient has been identified as being someone for whom the risk of blood clots is high, but for whom bleeding risk is estimated to be low.

The pop-up alert will be enabled in a sequential fashion for each group of hospitals in 1 month blocks. We will look to see if the pop-up alert changes the number of patients who receive rivaroxaban. We will also measure the outcomes of blood clots and bleeding among all discharging patients.

DETAILED DESCRIPTION:
The goal of this prospective, cluster, randomized, type II hybrid step wedge, implementation/effectiveness study is to compare the rates of rivaroxaban prescription for extended duration thromboprophylaxis (EDT) in discharging medical patients during the baseline period when no alert informs decision-making to guide EDT, versus EDT prescription during the intervention period when an alert to the discharging clinician is delivered.

Grouped sequential hospitals will be introduced to the intervention randomly in a step wedge fashion.

Aim 1 is to assess the implementation of the alert to discharging clinicians caring for eligible hospitalized medical patients. The primary outcome for Aim 1 is the comparative rate of prescription of EDT (rivaroxaban 10 mg daily for 30 days) during the baseline period versus the intervention period among eligible patients.

Secondary outcomes for Aim 1 will capture interactions with the alert.

Aim 2 is to assess the impact of the alert on important patient clinical outcomes.

The primary efficacy outcome for Aim 2 is the composite of 90-day venous thromboembolism, non-hemorrhagic stroke, myocardial infarction and death.

The primary safety outcome for Aim 2 is 30-day major bleeding. Secondary outcomes for Aim 2 will be the net clinical benefit, defined as the primary outcome + the primary safety outcome during the baseline phase versus the intervention phase among all at risk patients, and all patients for which an alert leads to the prescription of EDT.

Additional secondary outcomes will report components of the primary efficacy and safety outcomes in various groups.

ELIGIBILITY:
Inclusion Criteria:

* Discharging clinician must be in one of the following iCentra electronic health record (Cerner, Kansas City, MO) positions:

  * Physician, nurse practitioner, or physician assistant hospitalist
  * Physician internal medicine
  * Physician family medicine
* Patient age ≥ 18 years.
* The encounter must be inpatient.
* A signed hospital discharge order must be present.
* eVTE target population criteria (increased venous thromboembolism risk, low bleeding risk) must be met

Exclusion Criteria:

* Pregnant during encounter
* Discharge order completed by ineligible clinician type
* Exclude all cases where the patient is being actively prescribed and intended to be discharged on the following qualifying anticoagulant medications, regardless of dose form or dosing regimen (i.e., they have an active prescription for one of these medications):

  * Apixaban
  * Dabigatran
  * Dalteparin
  * Enoxaparin
  * Edoxaban
  * Betrixaban
  * Fondaparinux
  * Rivaroxaban
  * Warfarin
* Creatinine clearance <30 milliliters/minute based on last-available eligible serum creatinine value preceding discharge

  * Estimated creatine clearance based on actual body weight (preferred) ((140 - age years) * measured weight kilograms) / (72.0 * serum creatine milligrams/deciliter) (*0.85 if female)) = milliliters/minute
  * If measured body weight not available, then based on ideal body weight ((140 - age years) * ideal body weight kilograms) / (72.0 * serum creatine milligrams/deciliter) (*0.85 if female)) = milliliters/minute

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152000 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary outcome (implementation) | From discharge to 7 days after discharge
  Proportion of rivaroxaban prescriptions sent during the intervention phase, compared to the baseline phase
Primary clinical efficacy outcome (effectiveness) | From enrollment until 90 days after enrollment
  Composite of 90-day venous thromboembolism, myocardial infarction, non-hemorrhagic stroke, or death during the intervention phase for those patients for whom an alert was generated, compared to eligible at-risk patients during the baseline phase for whom no alert was generated
Primary clinical safety outcome | From enrollment until 30 days after enrollment
  30 day major bleeding during the intervention phase for those patients for whom an alert was generated and a prescription was sent, compared to eligible at-risk patients during the baseline phase for whom no alert was generated

CONTACTS AND LOCATIONS:
Overall Officials: Scott C. Woller, MD, Principal Investigator — Intermountain Health
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hyder SN, Han HB, Ash S, Horne BD, Stevens SM, Woller SC, Barnes GD. Predicting post-discharge venous thromboembolism and bleeding among medical patients: External validation of a novel risk score utilizing ubiquitous biomarkers. Thromb Res. 2023 Jul;227:45-50. doi: 10.1016/j.thromres.2023.05.011. Epub 2023 May 19. PMID 37235947
- [Background] Woller SC, Stevens SM, Bledsoe JR, Fazili M, Lloyd JF, Snow GL, Horne BD. Biomarker derived risk scores predict venous thromboembolism and major bleeding among patients with COVID-19. Res Pract Thromb Haemost. 2022 Jul 21;6(5):e12765. doi: 10.1002/rth2.12765. eCollection 2022 Jul. PMID 35873221
- [Background] Woller SC, Stevens SM, Fazili M, Lloyd JF, Wilson EL, Snow GL, Bledsoe JR, Horne BD. Post-discharge thrombosis and bleeding in medical patients: A novel risk score derived from ubiquitous biomarkers. Res Pract Thromb Haemost. 2021 Jul 7;5(5):e12560. doi: 10.1002/rth2.12560. eCollection 2021 Jul. PMID 34263106